CLINICAL TRIAL: NCT01720823
Title: Diagnostic Characteristics of a Home Polysomnograph for the Diagnosis of Patients With Obstructive Sleep Apnea Syndrome - A Pilot Study
Brief Title: Obstructive Sleep Apnea Syndrome (OSA) and Getemed
Acronym: GETEMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009.589
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea syndrome; polysomnography; Home monitoring
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- home polysomnography and standard polysomnography (Experimental): home polysomnography (GETEMED) and standard polysomnography (BRAINNETII) are both carried out in children during 1 night.
  Interventions: Device: home polysomnography (GETEMED); Device: standard polysomnography (BRAINNET II)

INTERVENTIONS:
Device: home polysomnography (GETEMED)
  Other Names: GETEMED
Device: standard polysomnography (BRAINNET II)
  Other Names: BRAINNET II

SUMMARY:
It is often clinically impossible to differentiate children with an isolated snoring from those with OSA. The diagnosis of OSA is currently based on nocturnal, laboratory-based polysomnography. This expensive examination is poorly accessible due to appointments delays at hospital.

Our study is designed to compare the characteristics of a home polysomnography versus standard polysomnography for the diagnosis of pediatric OSA.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 2 to 6 years old, requiring a polysomnography or admitted for intense snoring or suspected sleep apnea
* Parents must have signed the inform consent form and be covered by the National Health Insurance Program.

Exclusion Criteria:

* Parents opposed to the study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2012-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Characteristics of a home polysomnograph versus standard polysomnography for the diagnosis of OSA in children. | 1 night
  * Standard polysomnography considered pathological if obstructive apnea-hypopnea index (AHI) > 5 / hr.
  * Home polysomnography considered pathological if at least one of the following criteria is present :
    1. Respiratory Disturbance Index (RDI) > 10 / hr + /- Desaturation Index > 4% for more than 2.5 / hr.
    2. Brouillette index ; pulse wave > 3 desaturation clusters and > 3 desaturation <90%.

SECONDARY OUTCOMES:
To determine polygraphic pathological criteria by comparing the RDI per hour of the home polysomnography versus the (AHI) of the standard polysomnography. | 1 night

CONTACTS AND LOCATIONS:
Overall Officials: Patricia FRANCO, MD, Principal Investigator — Hospices Civils de Lyon- Hôpital Femme Mère Enfant
Locations (1):
- Hospices Civils de Lyon- Hôpital Femme Mère Enfant, Bron, France